CLINICAL TRIAL: NCT03840434
Title: COmpartment Syndrome vaLidation Of Non Invasive Assessment of Tissue Pressure (COLONIA)
Brief Title: COmpartment Syndrome vaLidation Of Non Invasive Assessment of Tissue Pressure
Acronym: COLONIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-A00141-56
Record Dates: First submitted 2019-01-28; First posted 2019-02-15 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Compartment Syndrome
Keywords: compartment syndrome; intramuscular punction Versus non invasive assessment
MeSH Terms: conditions — Compartment Syndromes

STUDY DESIGN:
Intervention Model Description: Each patient will perform a stress test to trigger the painful. Measurements will be done by intramuscular punction as usually, and by non invasive tool : MyotonPRO.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CCS group (Other): Measurements by intramuscular punction and non invasive tool
  Interventions: Diagnostic Test: MyotonPRO

INTERVENTIONS:
Diagnostic Test: MyotonPRO — Each patient will perform a stress test to trigger the painful. Measurements will be done by intramuscular punction as usually, and by non invasive tool : MyotonPRO

SUMMARY:
Chronic Compartment Syndrome (CCS) is a pathology that affects more specifically subjects exposed to repeated movements, particularly in a professional life or sports. The diagnosis is difficult and often delayed.

Currently, the reference technique is invasive. It consists of measuring by a intramuscular puncture (IMP) pressure in the offending compartment early after effort (usually between 1 and 5 minutes post-exercise). A value greater than or equal to 30 mmHg in the first 5 minutes is used as a diagnostic criterion for CCS.

Other less invasive techniques (scintigraphy) exist but are subject to certain discordances of interpretation. The advent of new assessment tools, like the MyotonPRO, pave the way for a non-invasive diagnostic approach.

DETAILED DESCRIPTION:
Patients referred for suspected chronic compartment syndrome causing will be included.

After signing the consent, the subject will have a clinical and paraclinical examination. Age, sex, height, weight, side of clinical symptomatology will be collected. Medical history current treatments will also be noted. Once the consent is collected, the patient performs, according to the data of the literature and service habits a stress test aimed at triggering the painful symptomatology associated with post-exercise IMP and MyotonPRO measurements as the same time.

ELIGIBILITY:
Inclusion Criteria:

* Affiliation to the French National healthcare system
* French speaking patients
* Referred for investigation of compartment syndrome causing

Exclusion Criteria:

* Pregnancy
* Inability to understand the study goal
* Patients protected by decision of law
* Extended dermatosis
* Coagulation disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-06-19 (Actual); Primary Completion 2023-03-27 (Actual); Study Completion 2023-03-27 (Actual)

PRIMARY OUTCOMES:
Diagnostic performance of MyotonPRO | 3 years
  To study the diagnostic performance of tissue stiffness measurement by MyotonPRO at 1 minute post-exercise in patients suspected of anterolateral of leg

SECONDARY OUTCOMES:
Diagnostic performance of MyotonPRO at 1 minute post-exercise | 3 years
  To study the diagnostic performance of the MyotonPRO tissue stiffness measurement variation between rest and 1 minute post-exercise.
Diagnostic performance of MyotonPRO at 5 minute post-exercise | 3 years
  To study the diagnostic performance of the MyotonPRO tissue stiffness measurement variation between rest and 5 minute post-exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Antoine BRUNEAU, PhD, Principal Investigator — UH Angers
Locations (1):
- Centre hospitalier universitaire, Angers, France

IPD SHARING:
Plan to Share IPD: Undecided